CLINICAL TRIAL: NCT03419923
Title: Three Anticoagulation Strategies for Hemodialysis in Patients at Risk of Hemorrhage: a Multicenter Randomized Trial
Brief Title: Three Anticoagulation Strategies for Hemodialysis in Patients at Risk of Hemorrhage
Acronym: TASHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GDREC2017250H
Record Dates: First submitted 2018-01-11; First posted 2018-02-05 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2017-12

CONDITIONS: Hemodialysis; Anticoagulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- saline flushes (Placebo Comparator): saline flushes with 250 mL were carried out every 30 min.
  Interventions: Drug: two stage regional citrate
- one stage regional citrate (Active Comparator): one stage regional citrate:4% trisodium citrate was infused at the arterial bubble trap at a rate according to the blood flow( 1.2 x blood flow)ml/h.
  Interventions: Drug: one stage regional citrate
- two stage regional citrate (Experimental): two stage regional citrate:4% trisodium citrate was infused at the arterial bubble trap at a rate according to the blood flow(3/4 x 1.2 x blood flow)ml/h,and at the venous bubble trap at a rate according to the blood flow(1/4 x 1.2 x blood flow)ml/h.
  Interventions: Drug: two stage regional citrate; Drug: one stage regional citrate

INTERVENTIONS:
Drug: two stage regional citrate — 4% trisodium citrate was infused at the arterial bubble trap at a rate according to the blood flow(3/4 x 1.2 x blood flow)ml/h,and at the venous bubble trap at a rate according to the blood flow(1/4 x 1.2 x blood flow)ml/h.
  Arms: saline flushes; two stage regional citrate
Drug: one stage regional citrate — 4% trisodium citrate was infused at the arterial bubble trap at a rate according to the blood flow( 1.2 x blood flow)ml/h.
  Arms: one stage regional citrate; two stage regional citrate

SUMMARY:
The aim of our study is to assess three anticoagulation strategies for intermittent hemodialysis(IHD) in patients at risk of hemorrhage. A registry of consecutive hemodialysis patients with high risk of hemorrhage was conducted at the Guangdong General Hospital, the First Affiliated Hospital of Guangzhou University of Chinese Medicine, the Second Affiliated Hospital of Guangzhou Medicine University or Guangzhou Hospital of Chinese Medicine, between Sep 10, 2017 and June 30th,2018. In this multi-center prospective and randomized study, participants were randomly divided into three groups during IHD according to different anticoagulation, including with regular saline flushes, one stage regional citrate anticoagulation (RCA) and two-stage RCA.

DETAILED DESCRIPTION:
Briefly, there are two parts in this study. The first part of the study is to compare two-stage RCA with one stage RCA during IHD, and the second part is to compare two-stage RCA with regular saline flushes, with estimated total procedures, 78 and 48, respectively. The primary outcome was measured as therapy interruption based on visible serious circuit clotting or persistent alarms such as venous pressure (> 200 mmHg) or TMP(transmembrane pressures) (> 300 mmHg). The secondary outcomes included circuit survival time, the total clotting score of ECC(extracorporeal circuit ) and urea clearance (Kt/V and URR). The total clotting score was the sum of the clotting scores for the venous expansion chamber, arterial expansion chamber, and dialyzer.

ELIGIBILITY:
Inclusion Criteria:

* age>=18 years
* intermittent hemodialysis patients that carry on a 4 hours hemodialysis procedure, 2-3 times one week.
* the therapy mode is hemodialysis，with a dialysis fluid more than 500ml/min and blood flow volume more than 3.5-4ml/min.kg；
* at risk of hemorrhage,including active hemorrhage(within 3 days),post-operation(within 3 days) and pre-invasive operation(within 7 days).

Exclusion Criteria:

* at high risk of citrate accumulation( total bilirubin >60umol/L; lactic acid>3mmol/L,）；
* use the drugs that impact the coagulation function within 7 days;
* serious hypocalcemia (serum calcium<1.9mmol/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2017-09-10 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
therapy interruption event | through study completion, from start to four hours
  visible serious circuit clotting or persistent alarms such as venous pressure (> 200 mmHg) or TMP (> 300 mmHg)dialyzer

SECONDARY OUTCOMES:
the clotting scores | through study procedure,an average of four hours
  the clotting scores in the venous expansion chamber, arterial expansion chamber and dialyzer
urea clearance | through study procedure,an average of four hours
  the measurement of Kt/V and URR

CONTACTS AND LOCATIONS:
Overall Officials: Liming Yao, M.D., Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593